CLINICAL TRIAL: NCT05512923
Title: Incidence and Risk Factors of Venous Thrombosis of the Lower Limbs After Hospitalization in Medical Patients at Risk
Acronym: MTE
Status: Recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Chef of Emergency Deparment, University of Monastir
Other Study IDs: MTE 2022
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Patients Hospitalized for More Than 48 Hours; Acute Medical Illness
Keywords: MTE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Tunisia, the available data are limited regarding the incidence of venous thrombosis of the lower limbs (TVMI) post-hospitalization, whether symptomatic or subclinical. The thromboprophylactic strategy will certainly depend on the incidence of this complication and its severity. In this study, we performed a systematic screening for TVMI in a well-characterized cohort of patients discharged after hospitalization >48h for an acute medical condition.

DETAILED DESCRIPTION:
This is a prospective follow-up of patients after hospitalization for more than 48 hours 6 weeks after discharge. The study must be approved by the ethics committee and all patients will have given their written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* patients included adults aged at least 40 years old
* hospitalized for more than 48 hours for an acute medical illness (i.e. heart failure, active cancer, acute ischemic stroke, infectious diseases, inflammatory disease and respiratory failure acute)
* patients at risk of MIVT due to moderate or severe immobility, history of thrombophilia (factor C or S deficiency, etc.), body mass index of 30 kg/m2.

Exclusion Criteria:

* hospitalised for less than 48
* patients who required intensive care, patients with cognitive impairment, patients admitted for SARS-CoV-2 infection or patients with a hospital stay <2 days, patients with a pre-existing reason for anticoagulation (therapeutic), such as atrial fibrillation or ETD and patients in whom MIVT is discovered on first ultrasound examination upon discharge from hospital.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients included adults aged at least 40 years old, hospitalized for more than 48 hours for an acute medical illness
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
presence of any symptoms suggestive of venous or arterial thromboembolic disease | Day7
  The first contact took place on day 7 after discharge from the hospital and is done by telephone. Patients will be asked about the presence of any symptoms suggestive of venous or arterial thromboembolic disease: angina, dyspnoea, peripheral edema, pain in the lower limbs or any other new symptom

SECONDARY OUTCOMES:
presence of any symptoms suggestive of venous or arterial thromboembolic disease | day45
  On D45, the patient will be seen again in the hospital. On the same day, the same symptoms will be sought and a second venous Doppler ultrasound of the lower limbs will be performed. If PE is suspected, a pulmonary CT angiography will also be performed.

CONTACTS AND LOCATIONS:
Overall Officials: nouira semir, Pr, Study Director — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- Nouira, Monastir, Tunisia